CLINICAL TRIAL: NCT05083741
Title: Head to Head Comparison of Chitodex Gel with Triamcinolone Vs NexFoam with Triamcinalone on Post-operative Outcomes in the Treatment of Chronic Rhinosinusitis (CRS)
Brief Title: Comparison of Chitodex Gel Vs NexFoam on Post-operative Outcomes in the Treatment of Chronic Rhinosinusitis
Status: Terminated | Type: Observational
Why Stopped: lack of recruitment and usable data
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Joseph Brunworth, MD, Assistant Professor, St. Louis University
Other Study IDs: 31454
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Chitogel: Chitodex gel plus Kenalog inserted into the middle meatus
  Interventions: Device: Chitogel
- Nexfoam: NexFoam plus Kenalog inserted into the middle meatus
  Interventions: Device: Nexfoam

INTERVENTIONS:
Device: Chitogel — post-operative dressing within standard of care
  Groups: Chitogel
Device: Nexfoam — post-operative dressing within standard of care
  Groups: Nexfoam

SUMMARY:
The purpose of this study is to compare the efficacy and outcomes of Chitodex gel plus Kenalog versus Nexfoam plus Kenalog in patients with chronic rhinosinusitis (CRS) undergoing sinus surgery. Both dressings are already known to be beneficial in controlling postoperative bleeding and promote wound healing.

DETAILED DESCRIPTION:
The trial will be single blinded randomized controlled trial and patients recruited will undergo endoscopic sinus surgery as standard of care for treatment of CRS. Specific outcome measures will be objective and subjective outcome scores post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Those who have had symptoms of chronic rhinosinusitis (nasal discharge, postnasal drip, nasal obstruction, facial pain and pressure, lack of sense of smell) that has been previously persistent for greater than 3 months AND
2. ≥ 18 years to ≤ 90 years AND
3. English speaking AND
4. Able to give written informed consent AND
5. Local residents who will be returning to this center for postoperative follow-up care AND
6. Indicated to undergo endoscopic sinus surgery and willing to return at 2-4, 6-8 & 12 (± 2) weeks post-op.

Exclusion Criteria:

1. allergy to shellfish
2. pregnant or breastfeeding
3. Hepatitis or blood disorders
4. any drug allergy
5. allergy to potato starch (due to Nexfoam)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SLUCare Otolaryngology Clinic
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Clinical Scores on Endoscopy | 12 (±2) weeks post surgery
  Outcome measured based on the wound healing in the sinus openings made during surgery.

SECONDARY OUTCOMES:
Symptom Scores on Patients' Self-Directed Questionnaires | 12 (±2) weeks post surgery
  Outcomes measured based on patients' personal symptom assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Brunworth, MD, Principal Investigator — Department of Otolaryngology-Head & Neck Surgery
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ngoc Ha T, Valentine R, Moratti S, Robinson S, Hanton L, Wormald PJ. A blinded randomized controlled trial evaluating the efficacy of chitosan gel on ostial stenosis following endoscopic sinus surgery. Int Forum Allergy Rhinol. 2013 Jul;3(7):573-80. doi: 10.1002/alr.21136. Epub 2013 Jan 16. PMID 23322408
- [Background] Le T, Psaltis A, Tan LW, Wormald PJ. The efficacy of topical antibiofilm agents in a sheep model of rhinosinusitis. Am J Rhinol. 2008 Nov-Dec;22(6):560-7. doi: 10.2500/ajr.2008.22.3232. PMID 19178792
- [Background] Jervis-Bardy J, Boase S, Psaltis A, Foreman A, Wormald PJ. A randomized trial of mupirocin sinonasal rinses versus saline in surgically recalcitrant staphylococcal chronic rhinosinusitis. Laryngoscope. 2012 Oct;122(10):2148-53. doi: 10.1002/lary.23486. Epub 2012 Aug 2. PMID 22865576